CLINICAL TRIAL: NCT07400445
Title: Interobserver Agreement Between Chest Radiograph and Computed Tomography for the Diagnosis of Acute Respiratory Distress Syndrome
Brief Title: Accuracy of the Chest Radiograph for the Diagnosis of Acute Respiratory Distress Syndrome
Acronym: CT 4 ARDS
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 29084890
Record Dates: First submitted 2026-01-30; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: acute respiratory distress syndrome; diagnostic imaging; computed tomography; chest radiograph; sensitivity; specificity
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The presence of bilateral lung infiltrates on chest imaging is a mandatory criterion for the diagnosis of acute respiratory distress syndrome (ARDS). This retrospective single-center observational study assessed the agreement between chest radiograph interpreted by intensivists and chest computed tomography interpreted by radiologists for the diagnosis of ARDS in mechanically ventilated patients with hypoxemia. Chest CT was considered the reference standard. The study evaluated interobserver agreement and diagnostic performance of chest radiography in the overall population and in predefined subgroups.

DETAILED DESCRIPTION:
Retrospective, single-center observational study conducted in the medical ICU of University Hospital of Poitiers, France, from January 1, 2015 to December 31, 2021. Included were intubated patients with PaO2/FiO2 ≤ 300 mmHg, PEEP ≥5 cmH2O, suspected ARDS except for imaging criterion, who underwent both chest CT and chest radiograph on the same day. Chest CT was interpreted by radiologists and used as reference for ARDS diagnosis. Chest radiographs were interpreted by intensivists. Agreement and diagnostic performance were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to intensive care unit
* Invasive mechanical ventilation
* Chest CT performed during ICU stay
* PaO2/FiO2 ≤ 300 mmHg with positive end-expiratory pressure ≥ 5 cmH2O the day of the CT-scan
* Chest radiograph performed within ± 24h of CT-scan

Exclusion Criteria:

* Cardiogenic pulmonary edema as the cause of hypoxemia
* Missing imaging data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the medical intensive care unit of the University Hospital of Poitiers
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Cohen's kappa coefficient for agreement between chest radiograph interpreted by intensivists and chest CT interpreted by radiologists for ARDS diagnosis. | Baseline
  0 indicates no agreement and 1 indicates perfect agreement

SECONDARY OUTCOMES:
Cohen's kappa coefficient for agreement between chest radiograph interpreted by intensivists and chest CT interpreted by radiologists for ARDS diagnosis in the subgroup of patients with moderate-to-severe hypoxemia | Baseline
  0 indicates no agreement and 1 indicates perfect agreement
Cohen's kappa coefficient for agreement between chest radiograph interpreted by intensivists and chest CT interpreted by radiologists for ARDS diagnosis in the subgroup of immunocompromised patients | Baseline
  0 indicates no agreement and 1 indicates perfect agreement
Cohen's kappa coefficient for agreement between chest radiograph interpreted by intensivists and chest CT interpreted by radiologists for ARDS diagnosis in the subgroup of obese patients | Baseline
  0 indicates no agreement and 1 indicates perfect agreement
Cohen's kappa coefficient for agreement between chest radiograph interpreted by intensivists and chest CT interpreted by radiologists for ARDS diagnosis in the subgroup of patients with 4 quadrants involved on chest radiograph | Baseline
  0 indicates no agreement and 1 indicates perfect agreement

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive Réanimation, University Hospital of Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable written request to the principal investigator, one year after publication of the main manuscript.
Time Frame: Start date: one year after publication of the main manuscript End date: two years after publication of the main manuscript